CLINICAL TRIAL: NCT05986162
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Preliminary Clinical Activity of Itolizumab in Subjects With Dermatomyositis
Brief Title: Safety and Preliminary Clinical Activity of Itolizumab in Dermatomyositis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BPL-ITO-DM-1001
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Dermatomyositis, Adult Type
MeSH Terms: conditions — Dermatomyositis | interventions — itolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Itolizumab Dose Level 1 (Experimental): Itolizumab of 25 mg administered by intravenous infusion every 2 weeks for a total of 7 doses.
  Interventions: Drug: Itolizumab
- Itolizumab Dose Level 2 (Experimental): Itolizumab of 50 mg administered by intravenous infusion every 2 weeks for a total of 7 doses.
  Interventions: Drug: Itolizumab
- Itolizumab Dose Level 3 (Experimental): Itolizumab of 100 mg administered by intravenous infusion every 2 weeks for a total of 7 doses.
  Interventions: Drug: Itolizumab

INTERVENTIONS:
Drug: Itolizumab — Patients to be treated with Itolizumab.
  Other Names: T1h

SUMMARY:
To evaluate the safety, tolerability, PK, PD, and preliminary clinical activity of Itolizumab in subjects with Dermatomyositis.

DETAILED DESCRIPTION:
The study will enroll approximately 44 subjects in two parts:

Part 1 is an open label, 3+3 single dose escalation and then mutiple dose administration phase. 9~30 patients with DM are expected to be enrolled across 3 dose cohorts.

Part 2 is a randomized phase and will enroll approximately 14 additional subjects, randomized in a 1:1 ratio to one of the 2 doses based on efficacy data obtained from Part 1. All participants in this study will receive Itolizumab intravenously every two weeks for a total of 7 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 18-75 years old (inclusive).
2. Fulfill one of the following criteria for DM:1) Bohan and Peter criteria for definite or probable DM;2) ENMC 2018 Dermatomyositis Classification Criteria
3. Disease activity fulfills at least three of the following criteria:1) MMT-8 score < 142; 2) physician's global disease activity ≥2 cm; 3) patient's global activity ≥2 cm; 4) extra-muscular activity ≥2 cm; 5) Health Assessment Questionnaire [HAQ] ≥0.25; 6) at least one muscle enzyme >1.5 times ULN
4. Under treatment with corticosteroids and/or at least 1 immunesuppressant, and being on stable therapy for at least 4 and 8 weeks for corticosteroids and immunesuppressant respectively (see Section 5.7.1)
5. Fulfill all of the following criteria: 1) % predicted values of FVC≥70%; 2) % predicted values of DLCO≥60%; 3) chest HRCT indicating the extent of disease lesion of DM-ILD < 20% as determined by the investigator
6. Negative result of serum HCG within 72 hours before enrollment for female with potential fertility
7. Able to understand and comply with the planned procedure as required by the protocol, and sign a written informed consent form (ICF)

Exclusion Criteria:

1. Subject with other connective tissue diseases (e.g., systemic sclerosis, systemic lupus erythematosus, rheumatoid arthritis, polyarteritis nodosa, Sjogren's syndrome, mixed connective tissue disease, etc.) or ANCA associated vasculitis.
2. Diagnosed with polymyositis or IMNM.
3. Diagnosed with systemic, severe musculoskeletal disorder that unrelated to DM and will interfere with the investigator's assessment of the subject's muscle strength.
4. Subject who plans to start a physical therapy program during the trial.
5. Subject who has a medical history of New York Heart Association class III or IV congestive heart failure, clinically significant or uncontrolled unstable angina or myocardial infarction, cerebrovascular accident, or pulmonary embolism within 6 months prior to screening
6. Subject with impaired renal function (serum creatinine > 1.5 x ULN or creatinine clearance < 30 mL/min [Cockcroft-Gault formula]) at screening.
7. Any of following significant abnormalities in liver function at screening:

   1. Serum alanine transaminase (ALT) or glutathione transaminase (AST) ≥ 3 x ULN, except when judged by the investigator to be due to DM;
   2. Total bilirubin ≥ 1.5 x ULN;
   3. Cirrhosis classification of Child-Pugh grade C.
8. Any of the following abnormalities at screening:

   1. Hepatitis B-related tests: ① positive hepatitis B surface antigen (HBsAg); ② positive hepatitis B core antibody (HBcAb); ③ positive hepatitis B surface antibody (HBsAb) and no history of hepatitis B vaccination; ④ positive hepatitis B e antigen or hepatitis B e antibody;
   2. Positive hepatitis C virus nucleic acid test (HCV-RNA);
   3. Positive acquired immunodeficiency syndrome antibody (HIV-Ab);
   4. Positive anti-syphilis spiral antibody (TP-Ab);
   5. Other acute or chronic infections requiring treatment.
9. Absolute lymphocyte count < 0.5×109/L at screening
10. Subject who has a medical history of tuberculosis or those who deny a history of tuberculosis but has a positive gamma-interferon release test at screening.
11. Any other clinically significant clinical condition or laboratory tests abnormality that, in the judgment of the investigator, may affect the safety evaluation
12. Any malignant tumor other than the cured carcinoma in situ or basal cell carcinoma within 5 years before screening
13. Suspected allergic to the investigational drug or any of its excipients
14. Subject who had participated in other clinical studies (other than those not receiving interventions, such as observational study or questionnaires survey) within 3 months prior to screening, or who are participating in other experimental treatments.
15. Subject who requires to be administrated with higher dose of corticosteroids and/or immunesuppressant than the allowed maximum dose specified in the protocol (section 5.7.1)
16. Subject who had been treated by one or more of the following drugs during the corresponding time window prior to screening:

    1. cyclophosphamide, rituximab within 12 months prior to screening;
    2. belizumab, tetrasip within 24 weeks prior to screening;
    3. intravenous immunoglobulin injections, baliximab, infliximab, adalimumab, tolimumab, JAK inhibitors within 12 weeks prior to screening;
    4. Other monoclonal antibodies or other biological agents within 12 weeks or 5 half-lives [whichever is longer] prior to screening.
17. Currently pregnant, breastfeeding,or planning to become pregnant or not using reliable method to avoid pregnancy during study and within 3 months after the last study treatment
18. As determined by the investigator, any medical, psychiatric, or other condition or circumstance that is likely to negatively affect the reliability of the study data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2025-05-03 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Study Week 20
  Number of subjects with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0

SECONDARY OUTCOMES:
Maximum serum concentration of Itolizumab, Cmax | Study Week 16
  Maximum serum concentration of Itolizumab
Minimum serum concentration of Itolizumab, Cmin | Study Week 16
  Minimum serum concentration of Itolizumab
Time to maximum serum concentration of Itolizumab, Tmax | Study Week 16
  Time to maximum serum concentration of Itolizumab
Total Itolizumab exposure across time, AUC0-t | Study Week 16
  Total Itolizumab exposure across time
Half life of Itolizumab, t1/2 | Study Week 16
  Half life of Itolizumab
IL-2 | Study Week 16
  Inflammatory Markers：IL-2
IL-6 | Study Week 16
  Inflammatory Markers:IL-6
TNF-α | Study Week 16
  Inflammatory Markers: TNF-α
IFN-γ | Study Week 16
  Inflammatory Markers:IFN-γ
CRP | Study Week 16
  Inflammatory Markers:CRP
Serum ferritin | Study Week 16
  Inflammatory Markers:Serum ferritin
ESR | Study Week 16
  Inflammatory Markers:ESR
IgG | Study Week 16
  Inflammatory Markers：IgG
IgM | Study Week 16
  Inflammatory Markers：IgM
IgA | Study Week 16
  Inflammatory Markers： IgA
CD6 receptor expression levels | Study Week 16
  Mean change of CD6 receptor expression levels in relative to baseline
T cell subsets | Study Week 16
  Mean change of different proportion of T cell subsets in relative to baseline
Proportion of patients achieving a TIS of ≥20 | Study Week 16
  Defined as patients with an increase of ≥20 points on the Total Improvement Score in relative to baseline.
Proportion of patients achieving DOI | Study Week 16
  DOI defined as ≥ 20% improvement in 3 of any 6 core set measures, with no more than 2 core set measures worsening by ≥ 25% (MMT-8 cannot worsen by ≥ 25%).
Mean Change of Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) activity score | Study Week 16
  Defined as the mean change of activity score of CDASI（Score Range：0~132，The hingher score indcates the worse outcome） relative to baseline.
Incidence of ADA | Study Week 16
  Defined as the precentage of subjects presenting anti-drug antibody

OTHER OUTCOMES:
Exploratory indicators | Study Week 16
  To explore wether the change of the antibody can indcates the clinical efficiency of Itolizumab in DM patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital; Rui Chen, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No